CLINICAL TRIAL: NCT05016180
Title: Impact of Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative Nausea and Vomiting and Early Outcome After Laparoscopic Bariatric Surgery: a Randomized Double-Blinded Controlled Trial
Brief Title: Effect of Ultrasound-guided Transversus Abdominis Plane Block After Laparoscopic Bariatric Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB2020-YX-083-01
Record Dates: First submitted 2021-06-30; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Nausea and Vomiting; Laparoscopic Bariatric Surgery
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): Before the induction of anesthesia, normal saline is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Ropivacaine
- Ropivacaine (Experimental): Before the induction of anesthesia, Ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Before the induction of anesthesia, ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side

SUMMARY:
Purpose:

To explore and compare Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative nausea and vomiting and Early Outcome After Laparoscopic Bariatric Surgery To evaluate and examine TAPB can reduce the application of intraoperative and postoperative opioids and the duration of analgesia

DETAILED DESCRIPTION:
Poor postoperative nausea and vomiting control is a leading factor that hinders the physical rehabilitation, and causes acute cognitive impairment and chronic pain syndrome. Recently, the multimodal analgesia strategies to minimise opioid-related side effects are highly desirable in open surgical procedures. The transversus abdominis plane block is a novel technique involving injection of local anaesthetic between the internal oblique and the transversus abdominis muscles of the abdominal wall. Although ropivacaine is most commonly used for this technique, the analgesic duration remains not dissatisfied. Herein, we will evaluate the efficacy of ultrasound-guided transversus abdominis plane (USG-TAP) block with ropivacaine in Laparoscopic Bariatric Surgery

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo Laparoscopic Bariatric Surgery
2. Subject's American Society of Anesthesiologists physical status is I-III.
3. BMI>35kg/m2
4. The subject's parent/legally authorized guardian has given written informed consent to participate

Exclusion Criteria:

1. Subject has a diagnosis of renal or liver failure.
2. Subject has a diagnosis of mental illness
3. Subject is allergy and contraindication to Ropivacaine.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre-existing therapy with opioids, intake of any analgesic drug within 48 hours before surgery.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Subject is pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-11-26 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | 72 hours after surgery
  Postoperative nausea and vomiting

SECONDARY OUTCOMES:
Cumulative Sufentanyl Consumption | 24 hours after surgery
  Each patient was administered analgesics using a PCA pump containing sufentanil (100μg) in normal saline at a total volume of 100 ml after leaving PACU. This device was set to deliver a basal infusion of 2 ml/h and bolus doses of 0.5 ml with a 15-min lockout period. Sufentanyl cumulative consumption is recorded 24 hours postoperatively
Time of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥4) is initially controlled by titration of sufentanyl
Occurrence of Side Effects | 24 hours after surgery
  Occurrence of side effects: nausea, vomiting, dizziness, headache, shivering, pruritus
Total Dose of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥4) is initially controlled by titration of sufentanyl.

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, Study Director — Tianjin Medical University General Hospital
Locations (2):
- China (2):
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Zhen Jia, Tianjin, Tianjin Municipality